CLINICAL TRIAL: NCT05025748
Title: Ask Questions (ASQ): Implementation of a Communication Intervention to Improve Patient-Oncologist Communication in the Outpatient Medical Oncology Setting
Brief Title: Ask Questions (ASQ):Implementation of a Communication Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Susan Eggly, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-025
Record Dates: First submitted 2021-08-02; First posted 2021-08-27 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Stage II Breast Cancer; Stage III Breast Cancer; Stage IV Breast Cancer; Stage II Colorectal Cancer; Stage III Colorectal Cancer; Stage IV Colorectal Cancer; Stage II Lung Cancer; Stage III Lung Cancer; Stage IV Lung Cancer; Stage II Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer; Stage II Ovarian Cancer; Stage III Ovarian Cancer; Stage IV Ovarian Cancer; Stage II Cervical Cancer; Stage III Cervical Cancer; Stage II Bladder Cancer; Stage III Bladder Cancer; Stage IV Bladder Cancer; Stage II Kidney Cancer; Stage III Kidney Cancer; Stage IV Kidney Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Urinary Bladder Neoplasms; Kidney Neoplasms | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health services research (ASQ brochure) (Experimental): Patients receive ASQ brochure and complete questionnaires over 30 minutes at baseline, over 10 minutes pre-clinic visit, and over 30 minutes post-clinic visit.
  Interventions: Behavioral: Behavioral Intervention

INTERVENTIONS:
Behavioral: Behavioral Intervention — Complete questionnaires
  Other Names: Questionnaire Administration

SUMMARY:
This clinical trial implements a communication intervention to improve patient-oncologist communication in the outpatient medical oncology setting. A communication brochure called the ASQ brochure may help patients prepare for the doctor visit by thinking through the questions that patients and patients' family want to ask the doctor.

DETAILED DESCRIPTION:
Patient-centered communication is critical to providing high-quality care. In patient-provider clinical interactions, providers are responsible for several aspects of patient-centered communication. However, to reach the goal of providing the best possible treatments, patients should also actively participate by asking questions and expressing their concerns. Question prompt lists, simple lists of questions provided to patients before clinic visits to help them prepare for the appointment, have been tested in several medical contexts and patient populations, including among an underserved, minority population in Detroit, and have been shown to contribute to improved outcomes related to better communication quality. Using a RE-AIM framework, this descriptive, mixed methods, single-arm intervention study assesses the implementation of an evidence-based communication intervention (question prompt list), the "ASQ brochure". The ASQ brochure is designed to improve patient-oncologist communication and other outcomes by improving patient self-efficacy for managing patient-physician interactions. Investigators will recruit 225 patients and implement the ASQ brochure at seven Karmanos Cancer Center network sites. Participants are newly diagnosed patients with (Stages I-IV) cancer for which systemic therapy is likely a recommended treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Have a first appointment to see a medical oncologist at a Karmanos Cancer Institute (KCC) site for medical/systemic treatment for a new, confirmed diagnosis of stages I-IV cancer
* Speak and read English well enough to be able to understand consent documents
* Given the diverse population seen at KCI, we will make attempts to recruit a representative sample. Our strategy will be simply to ask recruiters to make special attempts to recruit a representative sample. If that strategy fails after the first 10 patients we will build in requirements that at least 25% of the patients self-identify as non-White

Exclusion Criteria:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Self-efficacy in managing patient-physician interactions | Baseline (Time 1) to pre-clinic visit (TIme 2) post-clinic visit (TIme 3)
  20 items, 5-point Likert scale

SECONDARY OUTCOMES:
Change in knowledge related to the patient's cancer and treatment | Baseline (Time 1) to pre-clinic visit (TIme 2) post-clinic visit (TIme 3)
  6 investigator-developed questions; 5-point Likert scale (strongly disagree - strongly agree)
Change in trust in physicians | Baseline (Time 1) to post-clinic visit (Time 3)
  generally (before) and in a specific physician (after): (5 items20 Likert scale)
Change in distress | Baseline (Time 1) to pre-clinic visit (TIme 2) post-clinic visit (TIme 3)
  Distress thermometer (one item, Likert scale (no distress - extreme distress)
Perceptions of the Question Prompt List | Post-meeting (Time 3)
  10 items, 5-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Susan Eggly, PhD, Principal Investigator — Wayne State University
Locations (8):
- United States (8):
  - Karmanos Cancer Institute at McLaren Bay Region, Bay City, Michigan
  - Karmanos Cancer Institute at McLaren Clarkston, Clarkston, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute at McLaren Flint, Flint, Michigan
  - Karmanos Cancer Institute at McLaren Macomb, Mount Clemens, Michigan
  - Karmanos Cancer Institute at McLaren Central Michigan, Mount Pleasant, Michigan
  - Karmanos Cancer Institute at McLaren Northern Michigan, Petoskey, Michigan
  - Karmanos Cancer Institute at McLaren Port Huron, Port Huron, Michigan

IPD SHARING:
Plan to Share IPD: No